CLINICAL TRIAL: NCT01998698
Title: Monovision Correction Versus Multifocal Lens Insertion Following Emulsification Cataract Surgery
Brief Title: Monovision vs Multifocal Lens Insertion in Cataract Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Assistant Professor, Democritus University of Thrace
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 192/19-11-2013
Record Dates: First submitted 2013-11-19; First posted 2013-12-02 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Cataract
Keywords: cataract; phacoemulsification; monovision; multifocal lens
MeSH Terms: conditions — Cataract | interventions — visthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monovision Group (Active Comparator): Phacoemulsification surgery with intraocular lens implantation (monovision correction)
  Interventions: Procedure: Phacoemulsification surgery
- Multifocal Group (Active Comparator): Phacoemulsification surgery with intraocular lens implantation (multifocal lens insertion)
  Interventions: Procedure: Phacoemulsification surgery

INTERVENTIONS:
Procedure: Phacoemulsification surgery — Phacoemulsification surgery with intraocular lens implantation and monovision correction
  Other Names: Alcon Infiniti Vision System platform; Visthesia, Carl Zeiss, Germany; Alcon Intraocular lens SN60WF
  Arms: Monovision Group
Procedure: Phacoemulsification surgery — Phacoemulsification surgery with multifocal intraocular lens implantation
  Other Names: Alcon Infiniti Vision System platform; Visthesia, Carl Zeiss, Germany; Hoya Intraocular lens PY-60MV
  Arms: Multifocal Group

SUMMARY:
The investigators would like to assess whether monovision correction of multifocal lens insertion provides more satisfaction to cataract patients following an uncomplicated phacoemulsification surgery.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral senile cataract

Exclusion Criteria:

* Glaucoma
* Corneal pathology
* Fundus pathology
* Severe neurological/mental diseases that interfere with visual acuity
* Former intraocular operation

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
VF14 score | 6 months following operation

SECONDARY OUTCOMES:
Distant Visual Acuity | 6 months following surgery
Near Vision visual acuity | 6 months following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Principal Investigator — Assistant Professor
Locations (1):
- University Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece

REFERENCES:
- [Result] Labiris G, Giarmoukakis A, Patsiamanidi M, Papadopoulos Z, Kozobolis VP. Mini-monovision versus multifocal intraocular lens implantation. J Cataract Refract Surg. 2015 Jan;41(1):53-7. doi: 10.1016/j.jcrs.2014.06.015. Epub 2014 Jun 21. PMID 24962144